CLINICAL TRIAL: NCT04414306
Title: Screen to Save 2: Rural Cancer Screening Educational Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Judith R. Rees, Associate Professor, Department of Epidemiology, Geisel School of Medicine, Dartmouth College Associate Director for Community Outreach and Engagement, Norris Cotton Cancer Center, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D20038; P30CA023108-40S4 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Colorectal Cancer
Keywords: cancer; cancer screening; colorectal cancer; education; rural
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm 1 (Experimental): Participants who meet eligibility criteria will be able to enroll and participate on-line, with some participating in online or telephone survey follow-up.
  Interventions: Other: Online educational video and website module

INTERVENTIONS:
Other: Online educational video and website module — Participants will receive online education via a video and website. Key messages will include information on risk factors, prevention, screening recommendations, and screening options pertaining to colorectal cancer. Some participants will be asked to participate in three and/or six-month follow-up surveys administered online or by telephone.

SUMMARY:
The purpose of this study is to help the Dartmouth Cancer Center and the National Cancer Institute understand how to educate people about cancer screening.

DETAILED DESCRIPTION:
The Dartmouth Cancer Center's Community Outreach and Engagement Team will implement Screen to Save 2 using an online format. The education will be based on a set of key messages that cover information about colorectal cancer, including risk factors, prevention, screening recommendations, and screening options. Key messages provided by the National Cancer Institute will be tailored to the local context of NH and VT, including information about local options for getting screened for colorectal cancer.

Using online or telephone surveys, some participants will be contacted approximately three months after their initial participation. Some of the participants contacted after three months will again be contacted another three months later (six months after initial participation). The three- and six-month surveys will assess knowledge, attitudes, beliefs, and behaviors related to cancer screening, including outcomes from cancer screening.

The primary aim of the study is to implement and evaluate Screen to Save 2 outreach and educational activities to improve knowledge of colorectal cancer screening methods, to increase intent to get screened for colorectal cancer, and connect screening services to the target population.

ELIGIBILITY:
Inclusion Criteria:

* Resident of one of the RUCC 7-9 counties in New Hampshire or Vermont (Coos or Sullivan County, NH; Caledonia, Windsor, Windham, Orange, Orleans, Lamoille, or Essex County, VT) and
* Age 45-74 at the time of enrollment in the study

Exclusion Criteria:

- Cognitive impairment preventing participation in informed consent process

Three-Month Follow-Up Survey Inclusion Criteria:

A participant will be eligible for inclusion in the three-month follow-up survey if the participant completed the pre-test, educational intervention, and post-test and at the time of initial participation:

* Answered a colorectal cancer screening history question indicating that the participant has never received colorectal cancer screening OR does not know if he/she has received colorectal cancer screening previously OR
* Answered a series of questions indicating that the participant received prior colorectal cancer screening but may be overdue for colorectal cancer screening based on the type of colorectal cancer screening last reported and screening guidelines for the frequency of re-screening.

Six-Month Follow-Up Survey Inclusion Criteria:

A participant will be eligible for inclusion in the six-month follow-up survey if the participant participated in the three-month-follow up survey and at that time reported that having:

* A FIT/FOBT screening or Cologuard (stool) screening performed since the time of initial study participation, but having not received the results
* An abnormal FIT/FOBT, or Cologuard (stool) screening since the time of initial study participation, but had not received a diagnostic colonoscopy
* A colonoscopy since the time of initial study participation, but had not received the final results

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Rees, BM, BCh, MPH, PhD, Principal Investigator — Geisel School of Medicine, Dartmouth College
Locations (1):
- Dartmouth Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm 1
Started | 205
Completed | 205
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm 1
Number analyzed (Participants) | 205
Age, Customized [Count of Participants; unit: Participants]
  <55 | 40
  55-59 | 39
  60-64 | 57
  65-69 | 39
  70-74 | 30
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 165
  Man | 40
  Non-binary/gender nonconforming | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 202
  Other | 2
  Declined to Answer | 1
Region of Enrollment [Number; unit: participants]
  United States | 205
Educational attainment [Count of Participants; unit: Participants]
  High school diploma/GED or less | 11
  Some college | 39
  College graduate | 155
Number of Forms of Insurance [Count of Participants; unit: Participants]
  None | 2
  Single | 163
  Two or more | 40
Type of insurance [Count of Participants; unit: Participants]
  Current or former employer | 112
  Individual plan | 21
  Military | 8
  Medicare | 75
  Medicaid | 12
  Other | 18
Ever screened for CRC [Count of Participants; unit: Participants]
  Yes | 170
  No | 30
  I don't know | 5
Number of methods of CRC screening [Count of Participants; unit: Participants]
  Single method | 122
  Two or more methods | 48
  Never screened/don't know | 35
Type of CRC screening method [Count of Participants; unit: Participants]
  Colonoscopy | 158
  Sigmoidoscopy | 20
  FIT/FOBT | 25
  DNA (Cologuard) | 21
  Computed Tomography | 1
History of polyps [Count of Participants; unit: Participants]
  Yes | 71
  No | 115
  Data Missing | 19
History of CRC [Count of Participants; unit: Participants]
  Yes | 5
  No | 200
History of CRC in any first-degree relatives [Count of Participants; unit: Participants]
  Yes | 42
  No | 163
History of CRC in any distant relatives [Count of Participants; unit: Participants]
  Yes | 32
  No | 173

OUTCOME MEASURES:

1. Primary Outcome: Change in Correct Responses Regarding Knowledge Related to Colorectal Cancer Risk, Prevention, and Screening
Description: A pre-test and post-test are conducted with participants to assess changes in knowledge related to key learning outcomes expected from the educational intervention (assessed via 14 true/false and multiple-choice questions, reported as a percent change in points). An increased % change in points represents increased knowledge of each survey question and a value of 0 indicates knowledge did not change (a negative value would indicate decreased knowledge). % change is a unique number that was calculated as the difference between the % answering correctly after the intervention minus the % correct before the intervention; it is representative of the entire data set and not calculated on an individual participant level. P values (<0.05) are based on chi-square tests. Each row represents a unique survey question evaluating the topic listed in the row title.
Time Frame: pre-test administered immediately before educational intervention; post-test administered immediately after the educational intervention on day 1.
Measure: Number; unit: Percent Change
Arm/Group | Experimental Arm 1
Number analyzed (Participants) | 205
Percent Change
  Early detection improves outcome | -.5
  Role of polyps in the development of CRC | 0
  CRC can be asymptomatic | 1
  Where CRC starts in the body | 2
  What is Lynch Syndrome | 13
  Purpose of colonoscopy | 1
  Important not to skip screening if asymptomatic | -.5
  What the stool test checks for | 5
  Recommended age to start colonoscopy | 16
  Recommended age to start FIT/FOBT | 24
  Family history of CRC | .5
  Poor diet | 4
  Red and processed meats | 3
  Being overweight or obese | 7
  Tobacco use | 11
  Lack of physical activity | 18
  Heavy drinking | 19
  Role of physical activity in reducing CRC risk | 18
Statistical Analysis 1: Comparison: Experimental Arm 1; Change in knowledge for survey question "What is Lynch syndrome"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "Poor diet"; Test type: Other; p = .002, t-test, 2 sided
Statistical Analysis 3: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "red and processed meats"; Test type: Other; p = .048, t-test, 2 sided
Statistical Analysis 4: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "being overweight or obese"; Test type: Other; p = .008, t-test, 2 sided
Statistical Analysis 5: Comparison: Experimental Arm 1; Change in knowledge for "recommended age to start colonoscopy"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Experimental Arm 1; Change in knowledge for "Recommended age to start FIT/FOBT"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "tobacco use"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "lack of physical activity"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 9: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "heavy drinking"; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 10: Comparison: Experimental Arm 1; Change in knowledge related to risk factor "role of physical activity in reducing CRC risk"; Test type: Other; p < .0001, t-test, 2 sided

2. Primary Outcome: Change in Colorectal Cancer Screening and Other Risk Behavior Intentions
Description: A pre-test and post-test are conducted to assess behavioral intention related to five prevention and screening behaviors (assessed via 5 questions on a 5-point Likert scale: strongly agree (5), agree, unsure, disagree, strongly disagree(1). The values reported represent the difference between pre-intervention and post-intervention scores, calculated as a unique number for the total responding participants (not calculated individually). A positive change represents increased intent. Each row represents a unique survey question evaluating the topic listed in the row title.
Time Frame: pre-test administered immediately before educational intervention; post-test administered immediately after educational intervention on day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental Arm 1 Pre-Education; Experimental Arm 1 Post-Education: Participants who meet eligibility criteria will be able to enroll and participate on-line, with some participating in online or telephone survey follow-up.
  Online educational video and website module: Participants will receive online education via a video and website. Key messages will include information on risk factors, prevention, screening recommendations, and screening options pertaining to colorectal cancer. Some participants will be asked to participate in three and/or six-month follow-up surveys administered online or by telephone.
Arm/Group | Experimental Arm 1 Pre-Education | Experimental Arm 1 Post-Education
Number analyzed (Participants) | 205 | 205
score on a scale
  Get CRC screening | 4.54 (.68) | 4.66 (.59)
  Talk to a healthcare provider about CRC screening | 4.39 (.81) | 4.5 (.68)
  Eat healthier diet | 4.08 (.78) | 4.22 (.72)
  Increase physical activity | 4 (.8) | 4.2 (.71)
  Talk about CRC with family or friends | 3.89 (.9) | 4.15 (.84)
Statistical Analysis 1: Comparison: Experimental Arm 1 Pre-Education; Change in intention to get a CRC screening; Test type: Other; p = .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Experimental Arm 1 Pre-Education; Change in intention to talk to a healthcare provider about CRC screening; Test type: Other; p = .006, t-test, 2 sided
Statistical Analysis 3: Comparison: Experimental Arm 1 Pre-Education; Change in intention to talk to eat a healthier diet; Test type: Other; p = .0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Experimental Arm 1 Pre-Education; Change in intention to increase physical activity; Test type: Other; p < .0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Experimental Arm 1 Pre-Education; Change in intention to talk about CRC with family or friends; Test type: Other; p < .0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 day
Arm/Group | Experimental Arm 1
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 0/205
Other Adverse Events (participants affected / at risk) | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04414306/Prot_SAP_000.pdf